CLINICAL TRIAL: NCT00528112
Title: Multi-Center, Open-Label, Randomized Study to Assess the Safety and Contraceptive Efficacy of Two Doses ( in vitro12 µg/24h and 16 µg/24h) of the Ultra Low Dose Levonorgestrel Contraceptive Intrauterine Systems (LCS) for a Maximum of 3 Years in Women 18 to 35 Years of Age and an Extension Phase of the 16µg/24h Dose Group (LCS16 Arm) up to 5 Years
Brief Title: Levonorgestrel Contraceptive Intrauterine Systems (LCS) Pearl Index Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 91665; 310442 (Other: Company internal); G04209F (Other: Company internal); G04209G (Other: Company internal); 2007-000420-40 (EudraCT Number)
Record Dates: First submitted 2007-09-11; First posted 2007-09-12 (Estimated); Results first posted 2012-09-24 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2016-12

CONDITIONS: Contraception
Keywords: Contraception; Intrauterine; IUD; IUS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LCS12 (Experimental): Intrauterine levonorgestrel contraceptive system (LCS), releasing levonorgestrel (LNG) 12 microg/24 h in vitro
  Interventions: Drug: LCS12
- LCS16 (Experimental): Intrauterine levonorgestrel contraceptive system (LCS), releasing levonorgestrel (LNG) 16 microg/24 h in vitro
  Interventions: Drug: LCS16

INTERVENTIONS:
Drug: LCS12 — Intrauterine system (IUS) with Levonorgestrel, in vitro releasing rate 12 microg/24 h
  Arms: LCS12
Drug: LCS16 — Intrauterine system (IUS) with Levonorgestrel, in vitro releasing rate 16 microg/24 h
  Arms: LCS16

SUMMARY:
This is a study on a new low dose levonorgestrel contraceptive intrauterine systems (LCS). The purpose of the study is to investigate which of the 2 administered doses is the lowest effective intrauterine dose of Levonorgestrel (LNG) administered via the LCS for contraception during 3 years. The study was amended: the LCS16 arm will be extended up to 5 years

DETAILED DESCRIPTION:
Drop out-rate will be covered in Participant flow section.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 35 years (inclusive), in good general health and requesting contraception.
* Has regular menstrual cycles (length of cycle 21-35 days) (i.e., endogenous cyclicity without hormonal contraceptive use).

Exclusion Criteria:

* Known or suspected pregnancy or is lactating.
* History of ectopic pregnancies.
* Any genital infection (until successfully treated).
* Abnormal uterine bleeding of unknown origin.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2885 (Actual)
Dates: Start 2007-08; Primary Completion 2011-07 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (117):
- United States (50):
  - Mobile, Alabama
  - Glendale, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Carmichael, California
  - Pacific Palisades, California
  - San Diego, California
  - Torrance, California
  - Denver, Colorado
  - Littleton, Colorado
  - Boyton Beach, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Boise, Idaho
  - Idaho Falls, Idaho
  - Chicago, Illinois
  - Evansville, Indiana
  - South Bend, Indiana
  - Marrero, Louisiana
  - Boston, Massachusetts
  - Kalamazoo, Michigan
  - Chaska, Minnesota
  - Chesterfield, Missouri
  - Lincoln, Nebraska
  - Las Vegas, Nevada
  - Moorestown, New Jersey
  - New Brunswick, New Jersey
  - Albuquerque, New Mexico
  - New York, New York
  - New Bern, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Medford, Oregon
  - Portland, Oregon
  - Jenkintown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Columbia, South Carolina
  - Chattanooga, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Houston, Texas
  - Norfolk, Virginia
  - Seattle, Washington
  - Spokane, Washington
- Argentina (4):
  - Lanús Oeste, Buenos Aires
  - San Isidro, Buenos Aires
  - Buenos Aires, Ciudad Auton. de Buenos Aires
  - Rosario, Santa Fe Province
- Canada (10):
  - Calgary, Alberta
  - Winnipeg, Manitoba
  - Kingston, Ontario
  - London, Ontario
  - Waterloo, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Shawinigan, Quebec
  - Sherbrooke, Quebec
  - Saskatoon, Saskatchewan
- Santiago, Chile
- Finland (9):
  - Espoo
  - Helsinki
  - Joensuu
  - Kotka
  - Kuopio
  - Lahti
  - Oulu
  - Tampere
  - Turku
- France (8):
  - Compiègne
  - Grenoble
  - Le Chesnay
  - Lille
  - Nîmes
  - Quetigny
  - Reims
  - Roanne
- Hungary (8):
  - Szeged, Csongrád megye
  - Békéscsaba
  - Budapest
  - Eger
  - Esztergom
  - Kecskemét
  - Nyíregyháza
  - Szentes
- Mexico (5):
  - Torreón, Coahuila
  - México, D.F., Mexico City
  - Monterrey, Nuevo León
  - Hermosillo, Sonora
  - México, D.F.
- Netherlands (9):
  - Alkmaar
  - Eindhoven
  - Heerlen
  - Helmond
  - Hoofddorp
  - Nijmegen
  - Rotterdam
  - The Hague
  - Utrecht
- Norway (5):
  - Elverum
  - Kolbotn
  - Larvik
  - Oslo
  - Trondheim
- Sweden (8):
  - Gothenburg
  - Luleå
  - Malmo
  - Norrköping
  - Örebro
  - Stockholm
  - Umeå
  - Uppsala

REFERENCES:
- [Result] Nahum GG, Kaunitz AM, Rosen K, Schmelter T, Lynen R. Ovarian cysts: presence and persistence with use of a 13.5mg levonorgestrel-releasing intrauterine system. Contraception. 2015 May;91(5):412-7. doi: 10.1016/j.contraception.2015.01.021. Epub 2015 Feb 7. PMID 25661510
- [Result] Apter D, Gemzell-Danielsson K, Hauck B, Rosen K, Zurth C. Pharmacokinetics of two low-dose levonorgestrel-releasing intrauterine systems and effects on ovulation rate and cervical function: pooled analyses of phase II and III studies. Fertil Steril. 2014 Jun;101(6):1656-62.e1-4. doi: 10.1016/j.fertnstert.2014.03.004. Epub 2014 Apr 14. PMID 24726226
- [Result] Nelson A, Apter D, Hauck B, Schmelter T, Rybowski S, Rosen K, Gemzell-Danielsson K. Two low-dose levonorgestrel intrauterine contraceptive systems: a randomized controlled trial. Obstet Gynecol. 2013 Dec;122(6):1205-13. doi: 10.1097/AOG.0000000000000019. PMID 24240244
- [Derived] Gemzell-Danielsson K, Apter D, Hauck B, Schmelter T, Rybowski S, Rosen K, Nelson A. The Effect of Age, Parity and Body Mass Index on the Efficacy, Safety, Placement and User Satisfaction Associated With Two Low-Dose Levonorgestrel Intrauterine Contraceptive Systems: Subgroup Analyses of Data From a Phase III Trial. PLoS One. 2015 Sep 17;10(9):e0135309. doi: 10.1371/journal.pone.0135309. eCollection 2015. PMID 26378938
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Groups:
- LCS12: Intrauterine levonorgestrel contraceptive system (LCS), releasing levonorgestrel (LNG) 12 microg/24 h in vitro. Treatment up to 3 years.
- LCS16: Intrauterine levonorgestrel contraceptive system (LCS), releasing levonorgestrel (LNG) 16 microg/24 h in vitro. Treatment up to 5 years.
Period: Treatment up to 3 Years
Arm/Group | LCS12 | LCS16
Started | 1432 | 1453
Participants Received Treatment | 1432 (Full analysis set/Safety population) | 1452 (Full analysis set/Safety population)
Completed | 819 | 870
Not Completed | 613 | 583
Not completed — Adverse Event | 313 | 278
Not completed — Withdrawal by Subject | 26 | 31
Not completed — Protocol Violation | 16 | 16
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 63 | 61
Not completed — Pregnancy | 9 | 10
Not completed — Other reasons | 186 | 186
Period: Extension Phase
Arm/Group | LCS12 | LCS16
Started | 0 (Only subjects in the LCS16 groups could participate in the extension phase) | 707
Completed | 0 | 550
Not Completed | 0 | 157
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Other reasons | 0 | 100
Not completed — Pregnancy | 0 | 3
Not completed — Lost to Follow-up | 0 | 12
Not completed — Death | 0 | 1
Not completed — Adverse Event | 0 | 36
Not completed — Protocol Violation | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LCS12 | LCS16 | Total
Number analyzed (Participants) | 1432 | 1452 | 2884
Age, Continuous [Mean (Full Range); unit: Years] | 27.2 [18 to 35] | 27.1 [18 to 35] | 27.1 [18 to 35]
Age, Customized [Number; unit: Participants]
  ≤ 25 years | 566 | 564 | 1130
  > 25 years ≤ 35 years | 866 | 888 | 1754
Gender [Count of Participants; unit: Participants]
  Female | 1432 | 1452 | 2884
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pearl Index up to 3 Years
Description: The unadjusted Pearl Index (PI) is defined as the number of pregnancies per 100 woman years. The 3-year PI was obtained by dividing the number of pregnancies that occurred during the first three years of treatment by the time (in 100 women years) that the women were at risk of getting pregnant.
Time Frame: Up to 3 years
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: Pregnancies per 100 women years
Arm/Group | LCS12 | LCS16
Number analyzed (Participants) | 1432 | 1452
Pregnancies per 100 women years | 0.33 [0.16 to 0.60] | 0.31 [0.15 to 0.57]
Statistical Analysis 1: Comparison: LCS12; Cumulative failure rate (Kaplan-Meier) at 3 years; Test type: Superiority or Other; failure rate = 0.009, 95% CI 2-sided [0.005 to 0.017]
Statistical Analysis 2: Comparison: LCS16; Cumulative failure rate (Kaplan-Meier) at 3 years; Test type: Superiority or Other; failure rate = 0.010, 95% CI [0.005 to 0.018]

2. Secondary Outcome: Bleeding Patterns in Days by 90-day Reference Periods - Reference Period 1
Description: The occurrence of genital bleeding was to be recorded by study subjects every day in a diary. Bleeding was to be recorded as light, normal or heavy, no bleeding, or spotting only. Spotting was defined as slight genital bleeding relative to the participant's experience.
Time Frame: Day 1 to Day 90
Population: All participants from the full analysis set who had an assessment for this evaluation
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | LCS12 | LCS16
Number analyzed (Participants) | 1322 | 1348
Days
  Number of bleeding/spotting days | 40.9 (19.1) | 39.7 (19.2)
  Number of bleeding days | 18.3 (12.3) | 17.7 (13.2)
  Number of spotting only days | 22.6 (14.1) | 21.9 (14.0)

3. Secondary Outcome: Bleeding Patterns in Days by 90-day Reference Periods - Reference Period 2
Description: as for outcome 2
Time Frame: Day 91 to Day 180
Population: All participants from the full analysis set who had an assessment for this evaluation
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | LCS12 | LCS16
Number analyzed (Participants) | 1262 | 1300
Days
  Number of bleeding/spotting days | 23.3 (14.8) | 21.1 (15.1)
  Number of bleeding days | 10.2 (8.7) | 8.7 (9.1)
  Number of spotting only days | 13.2 (10.4) | 12.3 (10.4)

4. Secondary Outcome: Bleeding Patterns in Days by 90-day Reference Periods - Reference Period 3
Description: as for outcome 2
Time Frame: Day 181 to Day 270
Population: All participants from the full analysis set who had an assessment for this evaluation
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | LCS12 | LCS16
Number analyzed (Participants) | 1192 | 1238
Days
  Number of bleeding/spotting days | 19.4 (13.2) | 16.3 (12.8)
  Number of bleeding days | 8.3 (8.2) | 6.3 (7.5)
  Number of spotting only days | 11.2 (9.0) | 10.0 (8.8)

5. Secondary Outcome: Bleeding Patterns in Days by 90-day Reference Periods - Reference Period 4
Description: as for outcome 2
Time Frame: Day 271 to Day 360
Population: All participants from the full analysis set who had an assessment for this evaluation
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | LCS12 | LCS16
Number analyzed (Participants) | 1123 | 1175
Days
  Number of bleeding/spotting days | 17.6 (12.1) | 14.3 (11.8)
  Number of bleeding days | 7.2 (7.2) | 5.1 (6.6)
  Number of spotting only days | 10.4 (8.3) | 9.1 (8.2)

6. Secondary Outcome: Bleeding Patterns in Days by 90-day Reference Periods - Reference Period 12
Description: as for outcome 2
Time Frame: Day 991 to Day 1080
Population: All participants from the full analysis set who had an assessment for this evaluation
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | LCS12 | LCS16
Number analyzed (Participants) | 770 | 819
Days
  Number of bleeding/spotting days | 13.4 (9.9) | 10.2 (9.5)
  Number of bleeding days | 4.8 (5.9) | 3.3 (5.3)
  Number of spotting only days | 8.6 (7.1) | 6.9 (6.8)

7. Secondary Outcome: Bleeding Patterns in Days by 30-day Reference Periods - Reference Period 1
Description: as for outcome 2
Time Frame: Day 1 to Day 30
Population: All participants from the full analysis set who had an assessment for this evaluation
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | LCS12 | LCS16
Number analyzed (Participants) | 1355 | 1376
Days
  Number of bleeding/spotting days | 18.0 (8.0) | 17.3 (8.0)
  Number of bleeding days | 8.2 (6.0) | 8.1 (6.3)
  Number of spotting only days | 9.7 (6.5) | 9.2 (6.4)

8. Secondary Outcome: Bleeding Patterns in Days by 30-day Reference Periods - Reference Period 2
Description: as for outcome 2
Time Frame: Day 31 to Day 60
Population: All participants from the full analysis set who had an assessment for this evaluation
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | LCS12 | LCS16
Number analyzed (Participants) | 1345 | 1375
Days
  Number of bleeding/spotting days | 12.7 (7.6) | 12.9 (8.0)
  Number of bleeding days | 5.6 (4.9) | 5.5 (5.3)
  Number of spotting only days | 7.1 (5.9) | 7.3 (6.2)

9. Secondary Outcome: Bleeding Patterns in Days by 30-day Reference Periods - Reference Period 3
Description: as for outcome 2
Time Frame: Day 61 to Day 90
Population: All participants from the full analysis set who had an assessment for this evaluation
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | LCS12 | LCS16
Number analyzed (Participants) | 1328 | 1355
Days
  Number of bleeding/spotting days | 10.3 (6.9) | 9.5 (7.0)
  Number of bleeding days | 4.4 (4.1) | 4.1 (4.5)
  Number of spotting only days | 5.8 (5.2) | 5.4 (5.2)

10. Secondary Outcome: Bleeding Patterns in Days by 30-day Reference Periods - Reference Period 4
Description: as for outcome 2
Time Frame: Day 91 to Day 120
Population: All participants from the full analysis set who had an assessment for this evaluation
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | LCS12 | LCS16
Number analyzed (Participants) | 1300 | 1334
Days
  Number of bleeding/spotting days | 8.6 (6.0) | 7.8 (6.2)
  Number of bleeding days | 3.7 (3.6) | 3.2 (3.6)
  Number of spotting only days | 4.9 (4.5) | 4.6 (4.6)

11. Secondary Outcome: Bleeding Patterns in Days by 30-day Reference Periods - Reference Period 12
Description: as for outcome 2
Time Frame: Day 331 to Day 360
Population: All participants from the full analysis set who had an assessment for this evaluation
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | LCS12 | LCS16
Number analyzed (Participants) | 1130 | 1186
Days
  Number of bleeding/spotting days | 5.7 (4.7) | 4.6 (4.4)
  Number of bleeding days | 2.3 (2.8) | 1.6 (2.5)
  Number of spotting only days | 3.4 (3.4) | 3.0 (3.1)

12. Secondary Outcome: Number of Participants With/Without Ovulation - Year 1
Description: Serum concentrations of progesterone were analyzed. All subjects with progesterone values equal to or greater than 2.5 ng/ml were assessed as having an ovulation.
Time Frame: For six weeks in the second half of Year 1
Population: A subset of women from the full analysis set
Measure: Number; unit: Participants
Arm/Group | LCS12 | LCS16
Number analyzed (Participants) | 14 | 12
Participants
  With ovulation | 13 | 11
  Without ovulation | 1 | 1

13. Secondary Outcome: Number of Participants With/Without Ovulation - Year 2
Description: as for outcome 12
Time Frame: For six weeks in the second half of Year 2
Population: A subset of women from the full analysis set
Measure: Number; unit: Participants
Arm/Group | LCS12 | LCS16
Number analyzed (Participants) | 11 | 10
Participants
  With ovulation | 10 | 9
  Without ovulation | 1 | 1

14. Secondary Outcome: Number of Participants With/Without Ovulation - Year 3
Description: as for outcome 12
Time Frame: For six weeks in the second half of Year 3
Population: A subset of women from the full analysis set
Measure: Number; unit: Participants
Arm/Group | LCS12 | LCS16
Number analyzed (Participants) | 11 | 7
Participants
  With ovulation | 11 | 7
  Without ovulation | 0 | 0

15. Secondary Outcome: Average Total Cervical Score - Year 1
Description: Cervical mucus samples were analyzed to determine any effects of progesterone on the cervical mucus. Range of score: 0 (high contraceptive efficacy) to 12 (low contraceptive efficacy)
Time Frame: For six weeks in the second half of Year 1
Population: A subset of women from the full analysis set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | LCS12 | LCS16
Number analyzed (Participants) | 14 | 12
Scores on a scale | 3.067 (1.291) | 3.127 (1.620)

16. Secondary Outcome: Average Total Cervical Score - Year 2
Description: as for outcome 15
Time Frame: For six weeks in the second half of Year 2
Population: A subset of women from the full analysis set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | LCS12 | LCS16
Number analyzed (Participants) | 11 | 10
Scores on a scale | 3.358 (1.272) | 2.798 (1.499)

17. Secondary Outcome: Average Total Cervical Score - Year 3
Description: as for outcome 15
Time Frame: For six weeks in the second half of Year 3
Population: A subset of women from the full analysis set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | LCS12 | LCS16
Number analyzed (Participants) | 10 | 6
Scores on a scale | 2.837 (1.354) | 2.448 (1.521)

18. Secondary Outcome: Classification of Endometrium - Year 1
Description: The histological evaluation of the endometrium examined the effects of progesterone on the endometrium
Time Frame: At Year 1
Population: A subset of women from the full analysis set
Measure: Number; unit: Participants
Arm/Group | LCS12 | LCS16
Number analyzed (Participants) | 26 | 23
Participants
  Atrophic/inactive | 0 | 0
  Proliferative | 0 | 0
  Secretory | 25 | 22
  Menstrual | 0 | 0
  Unclassified | 1 | 1

19. Secondary Outcome: Classification of Endometrium - Year 2
Description: The histological evaluation of the endometrium examined the effects of progesterone on the endometrium
Time Frame: At Year 2
Population: A subset of women from the full analysis set
Measure: Number; unit: Participants
Arm/Group | LCS12 | LCS16
Number analyzed (Participants) | 22 | 19
Participants
  Atrophic/inactive | 0 | 0
  Proliferative | 0 | 0
  Secretory | 19 | 19
  Menstrual | 0 | 0
  Unclassified | 3 | 0

20. Secondary Outcome: Classification of Endometrium - Year 3 / End of Study
Description: The histological evaluation of the endometrium examined the effects of progesterone on the endometrium
Time Frame: At Year 3 / End of study
Population: A subset of women from the full analysis set
Measure: Number; unit: Participants
Arm/Group | LCS12 | LCS16
Number analyzed (Participants) | 25 | 23
Participants
  Atrophic/inactive | 0 | 0
  Proliferative | 0 | 1
  Secretory | 24 | 22
  Menstrual | 0 | 0
  Unclassified | 1 | 0

21. Secondary Outcome: Degree of User Overall Satisfaction With Study Treatment
Description: Overall user satisfaction was assessed by a questionnaire given to participants at the end of the study. The questionnaire was only given to participants whose end-of-study visit occurred after implementation of Protocol Amendment 3.
Time Frame: At the end of study/Year 3
Population: All participants from the full analysis set who had an assessment for this evaluation
Measure: Number; unit: Participants
Arm/Group | LCS12 | LCS16
Number analyzed (Participants) | 1053 | 1063
Participants
  Missing | 1 | 1
  Very satisfied | 796 | 842
  Somewhat satisfied | 201 | 177
  Neither satisfied / dissatisfied | 31 | 22
  Dissatisfied | 23 | 18
  Very dissatisfied | 1 | 3

22. Secondary Outcome: Number of Participants With Partial or Total Expulsion
Description: If LCS was displaced, but still in the cervical canal, it was assessed as being partially displaced. If LCS was expelled from the uterus, it was assessed as a total expulsion.
Time Frame: Up to 3 years
Population: All participants from the full analysis set who had an assessment for this evaluation
Measure: Number; unit: Participants
Arm/Group | LCS12 | LCS16
Number analyzed (Participants) | 1426 | 1445
Participants
  IUS partially expelled | 24 | 30
  IUS totally expelled | 29 | 16

23. Primary Outcome: Pearl Index for LCS16 up to 5 Years
Description: The unadjusted Pearl Index (PI) is defined as the number of pregnancies per 100 woman years.
Time Frame: Up to 5 years
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: Pregnancies per 100 women years
Arm/Group | LCS16
Number analyzed (Participants) | 1452
Pregnancies per 100 women years | 0.29 [0.16 to 0.50]
Statistical Analysis 1: Comparison: LCS16; Cumulative failure rate (Kaplan-Meier) at 5 years; Test type: Superiority or Other; failure rate = 0.01445, 95% CI 2-sided [0.00823 to 0.02531]

24. Secondary Outcome: Bleeding Patterns in Days by 90-day Reference Periods - Reference Period 13
Description: as for outcome 2
Time Frame: Day 1081 to Day 1170
Population: All participants from the full analysis set who had an assessment for this evaluation
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | LCS16
Number analyzed (Participants) | 617
Days
  Number of bleeding/spotting days | 9.6 (9.0)
  Number of bleeding days | 3.1 (4.8)
  Number of spotting only days | 6.6 (6.4)

25. Secondary Outcome: Bleeding Patterns in Days by 90-day Reference Periods - Reference Period 20
Description: as for outcome 2
Time Frame: Day 1711 to Day 1800
Population: All participants from the full analysis set who had an assessment for this evaluation
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | LCS16
Number analyzed (Participants) | 531
Days
  Number of bleeding/spotting days | 9.3 (8.8)
  Number of bleeding days | 2.9 (4.9)
  Number of spotting only days | 6.4 (6.1)

26. Secondary Outcome: Degree of User Overall Satisfaction With Study Treatment up to 5 Years
Description: as for outcome 21
Time Frame: At the end of study/Year 5
Population: All participants from the full analysis set who participated in the extension phase and had an assessment for this evaluation
Measure: Number; unit: Participants
Arm/Group | LCS16
Number analyzed (Participants) | 686
Participants
  Very satisfied | 610
  Somewhat satisfied | 70
  Neither satisfied / dissatisfied | 3
  Dissatisfied | 1
  Very dissatisfied | 2

27. Secondary Outcome: Number of Participants With Partial or Total Expulsion up to 5 Years
Description: as for outcome 22
Time Frame: Up to 5 years
Population: All participants from the full analysis set who had an assessment for this evaluation
Measure: Number; unit: Participants
Arm/Group | LCS16
Number analyzed (Participants) | 1445
Participants
  IUS partially expelled | 35
  IUS totally expelled | 19

ADVERSE EVENTS:
Time Frame: From start of treatment until end of study, up to 5 years.
Groups:
- LCS12, up to 3 Years: Intrauterine levonorgestrel contraceptive system (LCS), releasing levonorgestrel (LNG) 12 microg/24 h in vitro. Treatment up to 3 years.
- LCS16, up to 3 Years: Intrauterine levonorgestrel contraceptive system (LCS), releasing levonorgestrel (LNG) 16 microg/24 h in vitro. Treatment up to 3 years.
- LCS16, up to 5 Years: Intrauterine levonorgestrel contraceptive system (LCS), releasing levonorgestrel (LNG) 16 microg/24 h in vitro. Treatment up to 5 years.
Arm/Group | LCS12, up to 3 Years | LCS16, up to 3 Years | LCS16, up to 5 Years
Serious Adverse Events (participants affected / at risk) | 66/1432 | 72/1452 | 86/1452
Other Adverse Events (participants affected / at risk) | 952/1432 | 1014/1452 | 1054/1452
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCS12, up to 3 Years (N=1432) | LCS16, up to 3 Years (N=1452) | LCS16, up to 5 Years (N=1452)
Spherocytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0 | 0
Mitral valve prolapse (Cardiac disorders) | 0 | 1 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 1
Goitre (Endocrine disorders) | 1 | 1 | 1
Iridocyclitis (Eye disorders) | 1 | 0 | 0
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 4 | 4
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Salivary gland calculus (Gastrointestinal disorders) | 0 | 1 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Device dislocation (General disorders) | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 2 | 2
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 2 | 2
Gallbladder polyp (Hepatobiliary disorders) | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 6 | 7 | 8
Campylobacter gastroenteritis (Infections and infestations) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 1 | 1 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Genital herpes (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Meningitis (Infections and infestations) | 1 | 0 | 1
Meningitis viral (Infections and infestations) | 0 | 1 | 1
Pelvic inflammatory disease (Infections and infestations) | 2 | 4 | 5
Peritoneal abscess (Infections and infestations) | 1 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 1 | 1 | 1
Pneumonia (Infections and infestations) | 2 | 1 | 2
Pyelonephritis (Infections and infestations) | 1 | 1 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 2
Tonsillitis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0
Vestibular neuronitis (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 1
Streptococcal sepsis (Infections and infestations) | 1 | 0 | 0
Tubo-ovarian abscess (Infections and infestations) | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0
Herpes dermatitis (Infections and infestations) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Uterine perforation (Injury, poisoning and procedural complications) | 0 | 1 | 2
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 2 | 2
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 1
Weight increased (Investigations) | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Loose body in joint (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint instability (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 2
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Astrocytoma, low grade (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 2
Headache (Nervous system disorders) | 0 | 1 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1
Multiple sclerosis (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 1
Trigeminal neuralgia (Nervous system disorders) | 0 | 0 | 1
Status migrainosus (Nervous system disorders) | 1 | 0 | 0
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 3 | 0 | 0
Blighted ovum (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 | 6 | 7
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1
Affective disorder (Psychiatric disorders) | 0 | 1 | 1
Alcoholism (Psychiatric disorders) | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 1 | 1
Completed suicide (Psychiatric disorders) | 0 | 1 | 1
Depression (Psychiatric disorders) | 1 | 1 | 3
Depression suicidal (Psychiatric disorders) | 1 | 0 | 0
Drug dependence (Psychiatric disorders) | 0 | 1 | 1
Hallucination, auditory (Psychiatric disorders) | 1 | 0 | 0
Panic reaction (Psychiatric disorders) | 0 | 1 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
Polysubstance dependence (Psychiatric disorders) | 0 | 1 | 1
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Strangury (Renal and urinary disorders) | 1 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 2 | 2
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 | 1 | 1
Pelvic adhesions (Reproductive system and breast disorders) | 0 | 1 | 1
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0 | 0
Uterine spasm (Reproductive system and breast disorders) | 1 | 0 | 0
Ovarian cyst torsion (Reproductive system and breast disorders) | 0 | 1 | 1
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 2 | 0 | 0
Vaginal perforation (Reproductive system and breast disorders) | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Detoxification (Surgical and medical procedures) | 1 | 1 | 1
Hypertension (Vascular disorders) | 1 | 0 | 1
Varicose vein (Vascular disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCS12, up to 3 Years (N=1432) | LCS16, up to 3 Years (N=1452) | LCS16, up to 5 Years (N=1452)
Abdominal pain (Gastrointestinal disorders) | 96 | 98 | 102
Abdominal pain lower (Gastrointestinal disorders) | 67 | 62 | 74
Nausea (Gastrointestinal disorders) | 74 | 58 | 59
Influenza (Infections and infestations) | 72 | 92 | 100
Nasopharyngitis (Infections and infestations) | 103 | 109 | 122
Sinusitis (Infections and infestations) | 90 | 96 | 107
Urinary tract infection (Infections and infestations) | 156 | 148 | 167
Vaginal infection (Infections and infestations) | 48 | 62 | 73
Vulvovaginal candidiasis (Infections and infestations) | 72 | 74 | 86
Vaginitis bacterial (Infections and infestations) | 105 | 128 | 150
Vulvovaginal mycotic infection (Infections and infestations) | 99 | 108 | 126
Weight increased (Investigations) | 56 | 71 | 76
Back pain (Musculoskeletal and connective tissue disorders) | 59 | 65 | 80
Headache (Nervous system disorders) | 132 | 137 | 146
Cervical dysplasia (Reproductive system and breast disorders) | 107 | 116 | 147
Dysmenorrhoea (Reproductive system and breast disorders) | 130 | 109 | 116
Ovarian cyst (Reproductive system and breast disorders) | 186 | 303 | 337
Pelvic pain (Reproductive system and breast disorders) | 96 | 122 | 132
Vaginal haemorrhage (Reproductive system and breast disorders) | 66 | 73 | 80
Acne (Skin and subcutaneous tissue disorders) | 163 | 170 | 179

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal investigators (PIs) have to send the publication to sponsor 90 days prior to planned publishing. The sponsor has maximum 60 days for review and for recommending changes or mark parts that have to be deleted from the publication due to harming sponsor's confidentiality rights. Sponsor can request a delay in publication release up to 6 months.